CLINICAL TRIAL: NCT03008564
Title: Determining The Location and Ultrasound Anatomy of Two Previously Described Adductor Canal Block Approaches in Volunteers.
Brief Title: Adductor Canal Block Ultrasound Anatomy in Volunteers
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Yatish Siddapura Ranganath, Clinical Assistant Professor, University of Iowa
Other Study IDs: 201612345
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Adductor Canal Block; Postop Analgesia for Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Ultrasound scanning of the lower limb in volunteers — Several reference points will be marked by anatomical landmarks and/or ultrasound: the anterior superior iliac spine; base of patella; apex of the femoral triangle A measuring tape will be used to measure the anterior superior iliac spine (landmark); the base of the patella (landmark); apex of femoral triangle (ultrasound); and distal most portion of adductor canal (Point B described earlier; ultrasound). We will then measure the ASIS to: 1) base of patella; 2) apex of femoral triangle; and 3) Point B. We will repeat the same procedure on the opposite leg. Once complete, the volunteer will be allowed to dress and leave. The procedure should take approximately 10-20 minutes for each volunteer. The following things will be recorded for each subject:
  * Age
  * Gender
  * Weight
  * Height
  * BMI
  * Distance of ASIS to base of patella
  * Distance of Point A to base of patella
  * Distance of Point B to base of patella
  * Distance of apex of femoral triangle to base of patella

SUMMARY:
There has been dispute about the location at which the adductor canal block should be performed (3-6). Two Common approaches have been used for ultrasound guided adductor canal blocks with the 'point of entry' being:

1. Point A: midway point between the ASIS and base of patella
2. Point B: Point which is 2-3 cm proximal to the site where the femoral artery becomes the popliteal artery as it traverses away from the sartorius muscle towards the femur at the adductor hiatus (2)

We want to determine ultrasound anatomy in healthy volunteers by:

1. Measuring the distance between Point A and Point B
2. Studying the ultrasound anatomy at Point A and B - Determine their location with respect to the adductor canal and femoral triangle.

This will allow us to determine which is the best site for performing an adductor canal block

DETAILED DESCRIPTION:
It is important to answer the primary question because of the variable length of the adductor canal and we would like to determine the optimal position to perform the adductor canal block.

The adductor canal typically contains the saphenous nerve, nerve to vastus medialis muscle and on occasion, the obturator nerve (1). The roof of adductor canal is the vasto-adductor membrane and its length is reported to range from 5.5 cm to 15 cm with a mean of 7.6 cm2 and would suggest the length of the AC is variable. We would like to determine the length of the AC with the use of ultrasound. The AC would be determined to begin at the apex of the femoral triangle and end just proximal to the adductor hiatus. The length and location of the AC would be important to characterize as the volume of local anesthetic used and associated quadriceps weakness could be of significance in a shorter AC.

There has been dispute about the location at which the adductor canal block should be performed (3-6). Point A has been disputed to be within the femoral triangle and would therefore be a femoral nerve block as suggested by a small body of evidence (4-5). Clinically, it is unclear if there is a difference between quadriceps muscle weakness between the two approaches although it could be hypothesized placing a block at point A would lead to more quadriceps muscle weakness. With information gathered from this study, we plan to perform a clinical study by performing the nerve blocks at these two points with different volumes of local anesthetic and compare the amount analgesia and motor weakness between the two different approaches.

60 Volunteers (30 male and 30 female) aged between 18 to 75 years with a body mass index of 18 to 35 kg/m2 will be included in this study. Volunteers with previous surgery or deformities of the lower extremity will be excluded from the study

This is an observational study without a control group. Several reference points will be marked by anatomical landmarks and/or ultrasound:

A. the anterior superior iliac spine (landmark); B. the base of the patella (landmark); C. apex of femoral triangle (ultrasound); and D. distal most portion of adductor canal (Point B described earlier; ultrasound).

The primary outcome measure we are looking at is the distance between Point A and Point B.

We also plan to measure the distance (in centimeters) from:

1. Base of patella to Point A
2. Base of patella to Point B
3. Apex of the femoral triangle

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years, body mass index 18-35 kg/m2

Exclusion Criteria:

* no previous surgery or complaints from the lower extremity region

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We aim to recruit volunteers who principally are healthcare employees at UIHC who mainly work in the Main Operating Rooms and Ambulatory Surgical Center Operating Rooms, mainly due to ease of access to ultrasonographic equipment. The subjects include anesthesiologists, certified registered nurse anesthetists, residents, interns, nurses, volunteers, technicians, administrative staff and other members of staff working in these areas.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Measurement 1 | One time assessment done during Ultrasound scanning of the lower extremity
  The distance in cm between Point A and Point B

SECONDARY OUTCOMES:
Measurement 2 | One time assessment done during Ultrasound scanning of the lower extremity
  The distance in cm between Point A and base of patella
Measurement 3 | One time assessment done during Ultrasound scanning of the lower extremity
  The distance in cm between Point B and base of patella
Measurement 4 | One time assessment done during Ultrasound scanning of the lower extremity
  The distance in cm between Apex of femoral triangle and base of patella

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Yap, MBBS, Principal Investigator — 319-356-1616
Locations (1):
- University Of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bendtsen TF, Moriggl B, Chan V, Pedersen EM, Borglum J. Defining adductor canal block. Reg Anesth Pain Med. 2014 May-Jun;39(3):253-4. doi: 10.1097/AAP.0000000000000052. No abstract available. PMID 24747312
- [Background] Tubbs RS, Loukas M, Shoja MM, Apaydin N, Oakes WJ, Salter EG. Anatomy and potential clinical significance of the vastoadductor membrane. Surg Radiol Anat. 2007 Oct;29(7):569-73. doi: 10.1007/s00276-007-0230-4. Epub 2007 Jul 7. PMID 17618402
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Background] Bendtsen TF, Moriggl B, Chan V, Pedersen EM, Borglum J. Redefining the adductor canal block. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):442-3. doi: 10.1097/AAP.0000000000000119. No abstract available. PMID 25140514
- [Background] Bendtsen TF, Moriggl B, Chan V, Borglum J. Basic Topography of the Saphenous Nerve in the Femoral Triangle and the Adductor Canal. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):391-2. doi: 10.1097/AAP.0000000000000261. No abstract available. PMID 26079358
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251